CLINICAL TRIAL: NCT03140826
Title: Amplification and Selection of Antimicrobial Resistance in the Intestine II
Acronym: ASARI II
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Matthias Willmann, Prof. Dr. med., University Hospital Tuebingen
Other Study IDs: ASARI-II
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Antibiotic Selection Pressure
MeSH Terms: interventions — Meropenem; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Meropenem arm: Patients receiving meropenem to treat an infection.
  Interventions: Drug: meropenem
- Pip-Tazo arm: Patients receiving piperacillin-meropenem to treat an infection.

INTERVENTIONS:
Drug: meropenem — Antibiotics to treat infections.
  Other Names: piperacillin-tazobactam
  Groups: Meropenem arm

SUMMARY:
Stool samples will be collected from two groups of neutropenic patients in the case that a therapy with either meropenem or piperacillin/tazobactam is needed due to a suspected infection. The intestinal resistome will be determined and quantified using shotgun metagenomics. Based on this, regression models will be used to determine the actual selection pressure caused by these drugs, and both selective forces will be compared. The results will reveal if there is a drug that causes a lower selection pressure compared to the other. The study aims to generate knowledge that is required to design effective antibiotic stewardship programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemato-oncological disease in neutropenia or with expected neutropenia
* Need for treatment with meropenem or piperacillin-tazobactam

Exclusion Criteria:

* pregnancy
* HIV, HBV, HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemato-oncological disease in neutropenia or with expected neutropenia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic Selection Pressure | under treatment, max. 10 days
  Degree of the change of the intestinal resistome.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Willmann, Prof. Dr., Principal Investigator — University Tuebingen
Locations (2):
- Germany (2):
  - University Hospital Cologne, Cologne
  - Institute of Medical Microbiology and Hygiene, University Hospital of Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: No